CLINICAL TRIAL: NCT06347393
Title: Transgender and GENdEr diverSe Individuals Screening for Breast Cancer: the GENESIS Study
Brief Title: Transgender and Gender Diverse Individuals Screening for Breast Cancer
Acronym: GENESIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Istituto Europeo di Oncologia (Other); Luigi Sacco University Hospital (Other); Fatebenefratelli Hospital (Other); Ospedale Policlinico San Martino (Other); Università degli studi di Messina, Messina (Unknown); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Azienda USL Reggio Emilia - IRCCS (Other Government); Federico II University (Other); Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 6425
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography; Ultrasonography, Mammary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational Prospective Cohort (Other): Mammography and breast ultrasound
  Interventions: Diagnostic Test: Mammography and Breast Ultrasound

INTERVENTIONS:
Diagnostic Test: Mammography and Breast Ultrasound — Patients will be scanned using mammography and Breast Ultrasound for Breast Cancer Screening

SUMMARY:
The goal of this multicentric prospective study is to evaluate the incidence of Breast Cancer in transgender and gender-diverse population.

DETAILED DESCRIPTION:
In recent years, the scientific community has been paying increasing attention to lesbian, gay, bisexual, transgender, queer, intersexual, asexual population, with a special focus on transgender and gender-diverse individuals. Globally, the percentage of adults who identify themselves as transgender varies between 0.3% and 0.5%, while approximately 0.5% to 4.5% of adults are estimated to identify as gender-diverse. Despite the growing visibility of transgender and gender-diverse community and the efforts towards their depathologization, healthcare still needs to address two fundamental issues: the inadequate preparation of healthcare staff regarding gender incongruence which results in mistreatment and discrimination and the lack of uniform and large-scale prospective data. Scientific evidence regarding the risk of developing breast cancer (BC) in these patients and the related benefits of BC screening are still limited and insufficient. The Associazione Italiana di Oncologia Medica (AIOM), reported that the risk of developing BC tends to increase in transgender women compared to cisgender men (standardized incidence ratio [SIR], 46.7; 95% CI, 27.2-75.4), although it does not reach the level of risk in cisgender women (SIR, 0.3; 95% CI, 0.2-0.4). Conversely, in transgender men, the risk of BC decreases when compared to cisgender women (SIR, 0.2; 95% CI, 0.1-0.5), but it still remains higher than the risk present in cisgender men (58.9; 95% CI, 18.7-142.2).As for the screening programs, there is a lower adherence among the transgender and non-conforming-gender population compared to the cisgender population, due to socio-economic barriers and a lack of clear recommendations supported by scientific evidence.The National Comprehensive Cancer Network (NCCN)and AIOM guidelines currently do not include specific recommendations for transgender individuals due to the aforementioned lack of scientific evidence.

The American College of Radiology (ACR) regulates screening protocols for the transgender population based on factors such as age, hormone therapy exposure, surgical history, and risk categories.

ELIGIBILITY:
Inclusion Criteria:

* Transgender and gender-diverse individuals ≥18 years old who meet the ACR inclusion criteria
* Signed Informed Consent

Exclusion Criteria:

* Refuse to sign Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Breast Cancer | 1 year
  The incidence of BC in a selected population of transgender and gender-diverse individuals.

SECONDARY OUTCOMES:
The adherence rate to the screening | 1 year
  To evaluate the adherence rate to the screening, to estimate the relative risk of BC according to the subgroup of population considered and to identify risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Anna D'Angelo, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Advanced Radiology Center- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No